CLINICAL TRIAL: NCT04600466
Title: Identification of Molecular and Epidemiological Risk Factors in the Development of Gastric Cancer in High-risk Predominantly Hispanic Population
Brief Title: Molecular and Epidemiological Risk Factors in the Development of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: IIMS-UT Health San Antonio (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Mio Kitano, Clinical Investigator, The University of Texas Health Science Center at San Antonio
Other Study IDs: CTMS# 20-0084; KL2TR002646 (NIH); HSC20200467H (Other: University of Texas Health San Antonio)
Record Dates: First submitted 2020-10-09; First posted 2020-10-23 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Molecular Diagnostic Techniques; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — FFPE from gastric biopsy will be processed for molecular testing and retained for further testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Retrospective Non-Hispanics: Molecular testing will be done on formalin fixed paraffin-embeded (FFPE) tissue collected at the time of gastroadenocarcinoma diagnosis and subsequent biopsies. Participants who are alive will be asked to complete a survey and consent to germline testing.
  Interventions: Other: Molecular testing for all participants.; Other: Germline Testing; Other: Survey
- Retrospective Hispanic: Molecular testing will be done on formalin fixed paraffin-embeded (FFPE) tissue collected at the time of gastroadenocarcinoma diagnosis and subsequent biopsies. Participants who are alive will be asked to complete a survey and consent to germline testing.
  Interventions: Other: Molecular testing for all participants.; Other: Germline Testing; Other: Survey
- Prospective Non-Hispanic: Molecular testing will be done on formalin fixed paraffin-embeded (FFPE) tissue collected at the time of gastroadenocarcinoma diagnosis and subsequent biopsies. Participants will be asked to complete a survey and consent to germline testing.
  Interventions: Other: Molecular testing for all participants.; Other: Germline Testing; Other: Survey
- Prospective Hispanic: Molecular testing will be done on formalin fixed paraffin-embeded (FFPE) tissue collected at the time of gastroadenocarcinoma diagnosis and subsequent biopsies. Participants will be asked to complete a survey and consent to germline testing.
  Interventions: Other: Molecular testing for all participants.; Other: Germline Testing; Other: Survey

INTERVENTIONS:
Other: Molecular testing for all participants. — Molecular testing on formalin fixed paraffin-embedded (FFPE) tissues on retrospectively identified patients with gastric adenocarcinoma.
Other: Germline Testing — Germline testing will be done on prospectively identified patients and in retrospectively identified patients who are still alive.
Other: Survey — Survey will be administered on prospectively identified patients and in retrospectively identified patients who are still alive. Survey will be administered in person or via telephone. The survey in the language of the participants choice (English or Spanish) on sociodemographic information, current and/or prior PPI (proton pump inhibitor), H2 blocker, antibiotic, tobacco, alcohol, and recreational drug use. Questionnaire will include other risk factors for gastric adenocarcinoma such as certain dietary constituents (high salt diet, high consumption of processed meat, etc.) and occupational exposures.

SUMMARY:
This protocol is a single-institution feasibility study to identify the molecular and epidemiological risk factors in the development of gastric cancer in high-risk predominantly Hispanic South Texas population. The study is broken down into two main parts: 1) To identify molecular differences in gastric adenocarcinoma (GAC) between Non-Hispanics and Hispanics, stratified by age, and in benign, pre-malignant, and malignant gastric lesions; and 2) To identify environmental and clinicopathological factors in Hispanics associated with specific molecular changes linked to the development of GAC.

DETAILED DESCRIPTION:
The first part of the study will be accomplished by performing molecular testing on formalin-fixed paraffin-embedded (FFPE) tissues on retrospectively identified patients with GAC. Germline testing will be done on both retrospectively and prospectively identified cohort of patients with diagnosis of GAC. The second part of the study will be accomplished via survey administration on retrospectively and prospectively identified patients with diagnosis of GAC and to test Helicobacter pylori (H. pylori) and Epstein-Barr virus (EBV) infection status, which are known risk factors for the development of GAC, on their FFPE gastric specimen. The data from part 1 and part 2 will be analyzed and correlated. The overall goal of the study is to identify molecular markers and environmental risk factors in GAC unique to Hispanics relative to Non-Hispanics in South Texas, and to define molecular alterations in pre-malignant gastric lesions associated with the development of GAC. The long-term goal is to improve racial disparities by defining prognostic and therapeutic molecular markers and environmental risk factors in Hispanics and ultimately for all patients with GAC. Identification of high-risk molecular markers and environmental factors in the development of GAC will help future deployment of improved prevention and surveillance modalities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Patient with histologically confirmed diagnosis of gastric adenocarcinoma
* Able to understand English or Spanish (only for the prospective cohort)
* GEJ adenocarcinoma Type II (within 1 cm above and 2 cm below the GEJ) and Type III (2-5 cm below the GEJ)
* Hyperplastic polyps

Exclusion Criteria:

* Clinically AND genetically confirmed diagnosis of well-established hereditary cancer syndrome
* Gastroesophageal junction (GEJ) adenocarcinoma Type I (1-5 cm above the GEJ) as they are treated as esophageal cancer
* Other benign or malignant histology types (i.e. leiomyoma, gastrointestinal stroma tumors, fundic gland polyps, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of gastric adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2030-01-22 (Estimated); Study Completion 2030-01-22 (Estimated)

PRIMARY OUTCOMES:
To identify molecular differences in GAC between Non-Hispanics and Hispanics | 5 years
  DNA from archived FFPE gastric cancer tissue from patients with diagnosis of GAC will be analyzed for the top 25 mutated genes identified in The Cancer Genome Atlas. The results will be compared and analyzed between Hispanics and non-Hispanics. In addition, germline testing using a 156 gene panel using saliva will be performs on patients with GAC and compared between Hispanics and non-Hispanics. Difference in somatic and germline mutations will be analyzed in patients with GAC between Hispanics and non-Hispanics.
To identify molecular differences in GAC between benign, pre-malignant, and malignant gastric lesions | 5 years
  Archived FFPE slides will be separated into malignant, normal, and pre-malignant sections after histopathology review. These include normal or pre-malignant adjacent tissue from GAC specimen or from prior gastric biopsy specimen. FFPE samples will be stratified into 4 main groups: 1) normal/superficial gastritis (SG); 2) atrophic gastritis (AG)/intestinal metaplasia (IM); 3) dysplasia; and 4) gastric adenocarcinoma (GCA). Top genes among the 25 analyzed in Outcome 1 will be studied on 50 benign and 100 pre-malignant samples and compared to the results from GAC samples from Outcome 1.
To identify environmental and clinicopathological factors in Hispanics associated with specific molecular changes | 5 years
  A comprehensive survey will be administered to patients with diagnosis of GAC retrospectively (to those who are still alive) and prospectively to query their anthropomorphic data, medical co-morbidities, sociodemographic information, dietary constituents, and exposures to known risk factors in the development of GAC. FFPE with gastric cancer tissue will be tested for EBV and H. pylori retrospectively and prospectively to test for prior exposure to these infections that are known risk factors for GAC.

CONTACTS AND LOCATIONS:
Overall Officials: Mio Kitano, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States